CLINICAL TRIAL: NCT04455737
Title: Ex Vivo Intra-arterial Indigo Carmine Injection After Transanal Total Mesorectal Excision
Acronym: RLF
Status: Completed | Type: Observational
Sponsor: Walter Brunner (Other)
Responsible Party: Sponsor-Investigator, Walter Brunner, Senior Consultant, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: Chir202001; 2020-01324 (Other: Swissethics BASEC)
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Rectal Neoplasms
Keywords: indigo carmine; lymph node; pathology
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with indigo carmine stained specimen: Specimen which underwent pathologic work-up after ex vivo indigo carmine injection into the inferior mesenteric artery after transanal total mesorectal excision.
  Interventions: Other: injection of indigo carmine
- Patients with unstained specimen: Specimen which underwent pathologic work-up after transanal total mesorectal excision without indigo carmine dyeing.

INTERVENTIONS:
Other: injection of indigo carmine — Ex vivo intra-arterial injection of 20 ml indigo carmine solution (10mL, 0.4% indigo carmine with 10mL, 0.9% saline solution) in the transanal total mesorectal excision specimen via the inferior mesenteric artery.
  Groups: Patients with indigo carmine stained specimen

SUMMARY:
Background: An exact lymph node staging is essential in the treatment of rectal cancer.

Objective: The aim of this study was to assess the effect of indigo carmine injection on the number of retrieved and positive lymph nodes after transanal total mesorectal excision (taTME).

Design: This is a retrospective, non-randomised study. Settings: This study was conducted at a tertiary hospital by a multidisciplinary team.

Patients: Between 2013 and 2019, patients undergoing transanal total mesorectal excision were analysed. Patients with indigo carmine injection (intervention group) were compared to those without (control group).

Interventions: Transanal total mesorectal excision was performed with or without ex vivo intra-arterial indigo carmine injection.

Main Outcome Measures: The number of retrieved and positive lymph nodes was the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* elective, oncologic rectum resection in TaTME technique for proven or highly suspected rectal cancer.

Exclusion Criteria:

* abdominoperineal resection
* extended colon resection
* previous surgery of the rectum, the left colon or the mesocolon/-rectum
* patients rejecting retrospective data analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective, oncologic rectum resection in TaTME technique
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
retrieved lymph nodes | 1 - 7 days after surgery
  number of lymph nodes retrieved by pathologist from the specimen

SECONDARY OUTCOMES:
positive lymph nodes | 1 - 7 days after surgery
  number of lymph nodes with microscopic tumor infiltration
N stage | 1 - 7 days after surgery
  N stage according TNM version 7
survival | 5 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Walter Brunner, MD MSc MBA, Principal Investigator — Kantonsspital St. Gallen, Rorschach branch, Department of Surgery
Locations (1):
- Department of General, Visceral, Endocrine and Transplantation Surgery, Cantonal Hospital St. Gallen, Rorschach, Switzerland

IPD SHARING:
Plan to Share IPD: No